CLINICAL TRIAL: NCT01018563
Title: An Open Label Extension Study of the Efficacy of MORAb-003 in Subjects With Platinum-Sensitive Epithelial Ovarian Cancer in First Relapse
Brief Title: An Open Label Extension Study of the Efficacy of MORAb-003
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated by sponsor due to futile results in NCT00849667 study.
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-003-002A; 2009-015825-36 (EudraCT Number)
Record Dates: First submitted 2009-11-18; First posted 2009-11-23 (Estimated); Results first posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2015-11

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Extension study; Epithelial ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — farletuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- MORAb-003 (Experimental): Maintenance infusions of MORAb-003 every 3 weeks
  Interventions: Drug: MORAb-003

INTERVENTIONS:
Drug: MORAb-003 — Dose group to be determined by dose assigned in main study and patient's weight. Intravenous infusions are given every 3 weeks.
  Other Names: Farletuzumab

SUMMARY:
An open label extension of the MORAb-003-002 study in order to continue the active patients in the MORAb-003-002 study on maintenance MORAb-003 infusions after the main study is closed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed consent.
* Subjects must have been enrolled in and have met the inclusion/exclusion criteria of the MORAb-003-002 study.
* Subjects must have achieved a normalization of CA 125 levels and/or CR or PR (or stable disease and an investigator's assessment of a clinical benefit) after MORAb-003 in combination with standard chemotherapy and have not yet met the criteria for disease progression during participation in the MORAb-003-002 study.
* Subjects must be currently receiving single-agent MORAb-003 maintenance therapy.

Exclusion Criteria:

• Subjects that discontinued the MORAb-003-002 study for any reason.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-01-13 (Actual); Primary Completion 2013-03-05 (Actual); Study Completion 2013-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Weil, MD, Study Director — Morphotek
Locations (3):
- United States (2):
  - Sharp Memorial Hospital, Chula Vista, California
  - South Texas Oncology & Hematology, San Antonio, Texas
- Nationales Centrum fur Tumorerkrandungen, Heidelberg, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants participated and received single-agent farletuzumab maintenance therapy in MORAb-003-002 study (NCT00318370), achieved normalization of cancer antigen 125 levels and/or tumor assessment of complete/partial response(or stable disease and an investigator's assessment of a clinical benefit) after receiving farletuzumab plus chemotherapy to enter study.
Pre-assignment Details: Study enrolled 3 participants who participated in the MORAb-003-002 study (NCT00318370), achieved a normalization of CA 125 levels and/or complete response or partial response after MORAb-003 in combination with standard chemotherapy, and received single-agent MORAb-003 maintenance therapy.
Groups:
- Farletuzumab 62.5 mg/m^2: Participants received farletuzumab 62.5 milligram per meter square (mg/m^2), intravenous infusion once weekly at the same dose level which participants received in the MORAb-003-002 (NCT00318370) parent study for up to approximately 37.7 months in this study.
- Farletuzumab 100 mg/m^2: Participants received farletuzumab 100 mg/m^2, intravenous infusion once weekly at the same dose participants received in the MORAb-003-002 (NCT00318370) parent study up to approximately 37.7 months in this study.
Period: Overall Study
Arm/Group | Farletuzumab 62.5 mg/m^2 | Farletuzumab 100 mg/m^2
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Termination of the study by Sponsor | 2 | 1

BASELINE CHARACTERISTICS:
Population: As per the planned analysis, the intention to treat population analysis set included all 3 participants who were enrolled and received at least 1 dose of farletuzumab in this extension-of-treatment study.
Groups:
- Farletuzumab- All Participants: Participants received farletuzumab 62.5 or 100 mg/m^2, intravenous infusion once weekly at the same dose level which participants received in the MORAb-003-002 (NCT00318370) parent study for up to 37.7 months in this study.
Arm/Group | Farletuzumab- All Participants
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 58.0 [38 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Duration of Ovarian Tumor Marker (Cancer Antigen 125 [CA125]) Response
Description: The duration of CA125 response, was defined the time from the date of the initial CA125 response (i.e., prior to enrollment in the parent study, was the starting point for assessment) to the first documentation of progressive disease (PD) by either Gynecologic Cancer Inter Group (GCIG) criteria for CA125 level or by the date of death due to any cause, whichever occurred first. Disease progression per CA125 was defined as the first of 2 consecutive CA125 values greater than (>) twice the upper limit of normal (ULN) (i.e. 35 kilo unit per liter [kU/L]) on two occasions. C= data censored at earlier non-PD assessment if PD did not occur.
Time Frame: From screening of parent study (NCT00318370) until the current study was terminated (up to a maximum of 78.2 months including the parent study, or 37.7 months in this study only)
Population: Intent-to-treat population included all 3 participants who were enrolled. Data reported includes combined data from the parent study MORAb-003-002 (NCT00318370) and the current study MORAb-003-002A.
Measure: Number; unit: months
Groups:
- Farletuzumab 62.5 mg/m^2: Participants received farletuzumab 62.5 mg/m^2, intravenous infusion once weekly at the same dose level which participants received in the MORAb-003-002 (NCT00318370) parent study for up to approximately 37.7 months in this study.
- Farletuzumab 100 mg/m^2: Participants received farletuzumab 100 mg/m^2, intravenous infusion once weekly at the same dose which participants received in the MORAb-003-002 (NCT00318370) parent study for up to approximately 37.7 months in this study.
Arm/Group | Farletuzumab 62.5 mg/m^2 | Farletuzumab 100 mg/m^2
Number analyzed (Participants) | 2 | 1
months
  Participant 1 (dose group: 62.5 mg/m^2)-C: number analyzed (Participants) | 1 | 0
  Participant 1 (dose group: 62.5 mg/m^2)-C | 77.2 |
  Participant 2 (dose group: 62.5 mg/m^2)-C: number analyzed (Participants) | 1 | 0
  Participant 2 (dose group: 62.5 mg/m^2)-C | 73.3 |
  Participant 3 (dose group: 100 mg/m^2): number analyzed (Participants) | 0 | 1
  Participant 3 (dose group: 100 mg/m^2) |  | 18.0

2. Secondary Outcome: Progression-Free Survival (PFS) by GCIG
Description: PFS was defined as the time from the date of first dose of study medication during the parent study MORAb-003-002 (NCT00318370) to the date of disease progression (either by GCIG for CA125 criteria or standard RECIST v.1.0 criteria) or to the date of death due to any cause in this study. PD per CA125 was defined as the first of 2 consecutive CA125 values >2*ULN (35 kU/L) on two occasions. Participants who were alive with no disease progression were censored at either the date of last CA125 assessment or date of last objective tumor evaluation, whichever was later. PFS was also censored if a participant received a non-study anticancer therapy or procedure, with censoring occurring at the date of the last RECIST or CA125 assessment prior to the start of a non-study anticancer therapy or procedure (whichever was earlier). C= data censored at earlier non-PD assessment if PD did not occur.
Time Frame: From the first dose of study medication in the parent study (NCT00318370) until the current study was terminated (up to a maximum of 78.2 months including the parent study, or 37.7 months in this study only)
Population: as for outcome 1
Measure: Number; unit: months
Groups:
- Farletuzumab 62.5 mg/m^2: Participants received farletuzumab 62.5 mg/m^2, intravenous infusion once weekly at the same dose participants received in the MORAb-003-002 (NCT00318370) parent study up to approximately 37.7 months in this study.
Arm/Group | Farletuzumab 62.5 mg/m^2 | Farletuzumab 100 mg/m^2
Number analyzed (Participants) | 2 | 1
months
  Participant 1 (dose group: 62.5 mg/m^2)-C: GCIG: number analyzed (Participants) | 1 | 0
  Participant 1 (dose group: 62.5 mg/m^2)-C: GCIG | 77.8 |
  Participant 2 (dose group: 62.5 mg/m^2)-C: GCIG: number analyzed (Participants) | 1 | 0
  Participant 2 (dose group: 62.5 mg/m^2)-C: GCIG | 75.8 |
  Participant 3 (dose group: 100 mg/m^2): GCIG: number analyzed (Participants) | 0 | 1
  Participant 3 (dose group: 100 mg/m^2): GCIG |  | 25.1

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined from the date of first dose of farletuzumab during the parent study MORAb-003-002 (NCT00318370) to date of death due to any cause. Participants who were alive had their OS time censored at the date they were last known to be alive. C= data censored at date participant was last known to be alive.
Time Frame: From Baseline (Day 1) in the parent study (NCT00318370) until date of death from any cause in this study, or until the current study was terminated (up to a maximum of 78.2 months including the parent study, or 37.7 months in this study only)
Population: as for outcome 1
Measure: Number; unit: months
Arm/Group | Farletuzumab 62.5 mg/m^2 | Farletuzumab 100 mg/m^2
Number analyzed (Participants) | 2 | 1
months
  Participant 1 (dose group: 62.5 mg/m^2)-C: number analyzed (Participants) | 1 | 0
  Participant 1 (dose group: 62.5 mg/m^2)-C | 78.3 |
  Participant 2 (dose group: 62.5 mg/m^2)-C: number analyzed (Participants) | 1 | 0
  Participant 2 (dose group: 62.5 mg/m^2)-C | 76.7 |
  Participant 3 (dose group: 100 mg/m^2): number analyzed (Participants) | 0 | 1
  Participant 3 (dose group: 100 mg/m^2) |  | 59.5

4. Secondary Outcome: Duration of Second Remission
Description: The prolongation of second and subsequent responses to chemotherapy plus farletuzumab relative to initial remission was assessed. Length of first remission was determined in the parent study MORAb-003-002 (NCT00318370). The length of second remission (i.e., the first remission in this study) was calculated using the following formula: '(carboplatin/taxane start date in this study - carboplatin/taxane start date in NCT00318370 +1/30.4'. The length of second remission was censored at the date of study discontinuation if the participant did not receive any carboplatin/taxane therapy during this study. C = censored data.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: months
Groups:
- Farletuzumab 62.5 mg/m^2: Participants received chemotherapy plus farletuzumab 62.5 mg/m^2, intravenous infusion once weekly at the same dose participants received in the MORAb-003-002 (NCT00318370) parent study up to approximately 37.7 months in this study.
- Farletuzumab 100 mg/m^2: Participants received chemotherapy plus farletuzumab 100 mg/m^2, intravenous infusion once weekly at the same dose participants received in the MORAb-003-002 (NCT00318370) parent study up to approximately 37.7 months in this study.
Arm/Group | Farletuzumab 62.5 mg/m^2 | Farletuzumab 100 mg/m^2
Number analyzed (Participants) | 2 | 1
months
  Participant 1 (dose group: 62.5 mg/m^2): number analyzed (Participants) | 1 | 0
  Participant 1 (dose group: 62.5 mg/m^2) | 41.0 |
  Participant 2 (dose group: 62.5 mg/m^2)-C: number analyzed (Participants) | 1 | 0
  Participant 2 (dose group: 62.5 mg/m^2)-C | 74.2 |
  Participant 3 (dose group: 100 mg/m^2): number analyzed (Participants) | 0 | 1
  Participant 3 (dose group: 100 mg/m^2) |  | 29.5

5. Secondary Outcome: Duration of Third Remission
Description: The length of third remission (i.e., second remission in this study) was calculated using the following formula: '(subsequent carboplatin/taxane start date in this study - carboplatin/taxane start date in NCT00318370 +1)/30.4'. The length of third remission was censored at the date of study discontinuation if the participant did not receive subsequent chemotherapy (carboplatin/taxane) during this study. Censored data is reported for all participants.
Time Frame: From Baseline (Day 1) of this study until date of death from any cause, or until the study was terminated (up to a maximum of 37.7 months)
Population: Intent-to-treat population included all 3 participants who were enrolled. Here "overall number of participants analyzed" are participants who were available for this outcome measure.
Measure: Number; unit: months
Arm/Group | Farletuzumab 62.5 mg/m^2 | Farletuzumab 100 mg/m^2
Number analyzed (Participants) | 1 | 1
months | 37.3 | 25.0

6. Other Pre Specified Outcome: Number of Participants With Best Overall Response as Evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) V.1.0 Criteria
Description: Best overall response was the best response recorded from the start of treatment until disease progression/recurrence. Participants were assigned to one of the following categories of change in disease status: complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). CR was defined as CR in both target and non-target lesions with no new lesions. PR was defined as CR in target lesions and incomplete response or SD in non-target lesions with no new lesions, or PR in target lesions and non-PD in non-target lesions with no new lesions. SD was defined as SD in target lesions and non-PD in non-target lesions with no new lesions. PD was defined as PD in target lesions, any non-target lesions with either absence or presence of new lesions, or any target lesions, PD in non-target lesions with either absence or presence of new lesions, or any target or non-target lesions with new lesions.
Time Frame: From the start of the treatment until disease progression/recurrence (up to approximately 37.7 months)
Population: Intent-to-treat population included all 3 participants who were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Farletuzumab 62.5 mg/m^2 | Farletuzumab 100 mg/m^2
Number analyzed (Participants) | 2 | 1
Participants
  CR | 1 | 1
  SD | 1 | 0

ADVERSE EVENTS:
Time Frame: For each participant, from the first dose till 30 days after the last dose or up to study completion (approximately 37.7 months)
Description: Intention to treat population analysis set included all 3 participants who were enrolled.
Arm/Group | Farletuzumab 62.5 mg/m^2 | Farletuzumab 100 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Farletuzumab 62.5 mg/m^2 (N=2) | Farletuzumab 100 mg/m^2 (N=1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Farletuzumab 62.5 mg/m^2 (N=2) | Farletuzumab 100 mg/m^2 (N=1)
Hypertension (Vascular disorders) | 0 (0) | 1 (5)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (11)
Asthenia (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (4)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (4) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (93) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (3)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (7)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (3)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (3)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated by sponsor due to futile results in the NCT00849667 (MORAb003-004) study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other